CLINICAL TRIAL: NCT01704638
Title: Kinetics of Fluvoxamine and Digoxin in Subjects With Different MDR1 Genotypes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Sparve, MD, specialist in clinical pharmacology, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: fluvoxaminedigoxin
Record Dates: First submitted 2012-09-21; First posted 2012-10-11 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Fluvoxamine; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2677TT (Experimental): Plasma kinetics of fluvoxamine and digoxin in this genotype
  Interventions: Drug: fluvoxamine; Drug: Digoxin
- 2677GG (Other): plasma kinetics of fluvoxamine and digoxin in this genotype
  Interventions: Drug: fluvoxamine; Drug: Digoxin

INTERVENTIONS:
Drug: fluvoxamine
Drug: Digoxin

SUMMARY:
The investigators will compare plasma kinetics of two marker drugs in individuals with different genetic variations in the MDR1-gene. The hypothesis is that one group will have higher exposure than the other.

ELIGIBILITY:
Inclusion Criteria:

* - Healthy volunteer ≥ 18 years of age
* Normal kidney function as measured by GFR according to Cockroft-Gault (70-120 ml/min)
* Normal P-potassiumvalue (3,6-4,6 mmol/L)
* HF>50 and no AV-block on resting ECG. No other significant abnormalities as judged by the investigator.
* Subject giving written informed consent
* Subject capable of understanding instructions

Exclusion Criteria:

* - Pregnancy
* Ongoing infection
* Intake of medication, including natural remedies (for example St John´s wort), within one month prior to starting study except for paracetamol.
* Active drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Cmax of fluvoxamine and of digoxin | 2 days for fluvoxamine and 2 days for digoxin. Washout period of at least 1 week between the both parts. Total study time maximum 4 weeks.
  The participants are administered a single dose of fluvoxamine or digoxin. Plasma kinetics of fluvoxamine are followed for 36 hours. Plasma kinetics of digoxin are followed for 48 hours. There is a washout period between the both parts.

CONTACTS AND LOCATIONS:
Locations (1):
- CPTU, Stockholm, Sweden